CLINICAL TRIAL: NCT04521439
Title: Hybrid PET/MR Imaging to Assess Demyelination and Axonal Injury in Multiple Sclerosis
Brief Title: Accurate Diagnosis of Multiple Sclerosis Using PET/MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: (2020)CER(126)
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS Patients Group (Experimental)
  Interventions: Diagnostic Test: 18F-florbetapir PET+MRSI
- Healthy Volunteers Group (Sham Comparator)
  Interventions: Diagnostic Test: 18F-florbetapir PET+MRSI

INTERVENTIONS:
Diagnostic Test: 18F-florbetapir PET+MRSI — PET and MRS quantitative parameters in MS lesions are simultaneously analyzed using hybrid PET/MR for obtaining demyelination and neuronal damage information.

SUMMARY:
Multiple sclerosis (MS) is an immune-mediated chronic inflammatory demyelinating disease of the central nervous system. Its main feature is progressive demyelination, which ultimately leads to axon damage and neuron loss. MR is the main imaging technique in the current diagnostic criteria of MS. The conventional MR sequence recommended in this diagnostic criteria has high sensitivity for detecting demyelination and axon damage, but has poor specificity, which makes disease modification therapy (DMT) blind, and it is also difficult to accurately determine the long-term prognosis.

PET is a non-invasive molecular imaging technology that can quantitatively monitor physiological or pathological processes in vivo. 18F-labeled thioflavin derivative probe (18F-florbetapir) can bind to myelin basic protein in the white matter, providing quantitative assessment of myelin content. Our preliminary studies have confirmed that the uptake of 18F-florbetapir in MS lesions is significantly related to the myelin content measured by histological staining. Therefore, 18F-florbetapir PET may be a very effective myelin imaging technology.

Advanced MR sequence such as magnetic resonance spectroscopy (MRS) can evaluate axonal damage by analyzing neuronal activity marker N-acetyl aspartate (NAA). The new whole-brain fast 3D MRS sequence breaks through the bottleneck of low signal-to-noise ratio and spatial resolution of the current MRS sequence, and provides a reliable method for obtaining neuronal activity markers in the three-dimensional space of MS sporadic lesions in the whole brain.

Integrated PET/MR makes PET detector implant in the MR magnet, which realizes the simultaneous acquisition of PET and MR in one scan, ensuring the high consistency of the two modes. This makes it possible to simultaneously analyze PET and MRS quantitative parameters in multiple and different sizes of MS lesions, that is, to obtain two different pathological features of demyelination and neuronal damage. Separating these two pathological changes will help to more accurately and quantitatively evaluate the efficacy of DMT, program selection and prognostic judgment.

This project intends to recruit 30 MS patients between 18-65 years old, and 30 healthy volunteers with matched age and sex as normal controls. PET/MR imaging, serological examination and cerebrospinal fluid testing and scale evaluation will be performed. The aim of this project is to planned to establish a new imaging evaluation technology for accurate diagnosis and prognosis evaluation of MS.

ELIGIBILITY:
MS Patients Group:

Inclusion Criteria:

* between 18-65 years old;
* diagnosed with mild or moderate disease (EDSS score ≤ 5 points); it meets the 2017 new version of McDonald diagnostic criteria for multiple sclerosis.
* meet the diagnostic criteria of clinically isolated syndromes (CIS)

Exclusion Criteria:

* No brain surgery/no brain trauma/no history of brain disease (stroke), no other independent neurological or psychiatric history;
* No severe depression symptoms;
* No alcoholism or drug dependence (addiction);
* No other conditions that affect the smooth progress of the inspection: such as hearing impairment, comprehension impairment, poor compliance, etc.;
* No rheumatic diseases and other acute or chronic inflammations (required for hematological markers).
* No MR contrast agent allergy

Healthy Volunteers Group:

Inclusion Criteria:

* between 18-65 years old;
* able to understand the purpose of clinical research and test plan;
* In the brain MR assessment, it is judged as "normal (corresponding to age)"

Exclusion Criteria:

* Any major mental illness; history of schizophrenia or schizoaffective disorder
* Any important neurological disease, such as cerebrovascular disease, inflammation or infectious disease, demyelinating disease, neurodegenerative disease, history of epilepsy or history of physical or craniocerebral trauma or brain surgery or intracranial hematoma with permanent brain history of injury;
* Brain MR has pathological manifestations;
* Any major diseases or unstable conditions (such as unstable angina, myocardial infarction or coronary revascularization within 12 months before enrollment, heart failure, chronic renal failure, chronic liver disease, severe lung disease, blood disease, poorly controlled diabetes, chronic infections);
* Medical history of tumors (except skin or prostate cancer in situ) within 5 years before screening;
* High risk of drug allergy (such as patients with allergic asthma) or history of severe allergic reactions to allergens;
* History of alcohol or drug abuse/dependence;
* MR contraindications (such as pacemaker or nerve stimulator or metal foreign body, high fever, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Distribution Volume Ratio (DVR) | Baseline
  Dynamic parameter of 18F-florbetapir distribution for quantitatively assessing the demyelination
Change from Baseline DVR at 6 months | 6 months after baseline
  Change of 18F-florbetapir distribution in the demyelinated lesions after 6 months
Change from Baseline DVR at 1 year | 1 year after baseline
  Change of 18F-florbetapir distribution in the demyelinated lesions after 1 year
Standardized Uptake Value Ratio (SUVR) | Baseline
  Static parameter of 18F-florbetapir uptake for quantitatively assessing the demyelination
Change from Baseline SUVR at 6 months | 6 months after baseline
  Change of 18F-florbetapir uptake in the demyelinated lesions after 6 months
Change from Baseline SUVR at 1 year | 1 year after baseline
  Change of 18F-florbetapir uptake in the demyelinated lesions after 1 year
N-acetyl aspartate (NAA) quantification | Baseline
  Neuronal activity marker based on magnetic resonance spectroscopy imaging (MRSI)
Change from Baseline NAA at 6 months | 6 months after baseline
  Change of neuronal activity marker in the demyelinated lesions after 6 months
Change from Baseline NAA at 1 year | 1 year after baseline
  Change of neuronal activity marker in the demyelinated lesions after 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China